CLINICAL TRIAL: NCT03032887
Title: Reducing Visitors- and Personnel-associated Infection Risk by Special Agitation Incl. Voice Prompts for Hand Disinfection on Perinatal Care Stations
Brief Title: Reducing Visitors- and Personnel-associated Infection Risk on Perinatal Care Station
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Gregor Seliger, Chief resident, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Hygienic voice
Record Dates: First submitted 2017-01-17; First posted 2017-01-26 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hygiene
Keywords: hygiene; prenatal care; postnatal care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- voice prompts (Experimental): Agitation (education, reminders and optimising materials) plus voice prompts
  Interventions: Behavioral: voice prompts; Behavioral: agitation
- no voice prompts (Other): only Agitation (education, reminders and optimising materials); no voice prompts
  Interventions: Behavioral: agitation

INTERVENTIONS:
Behavioral: voice prompts — voice prompts on disinfectant dispenser
  Arms: voice prompts
Behavioral: agitation — Education, reminders and optimising materials

SUMMARY:
The rate of infectious diseases (amnioninfection syndrome (AIS), fetal inflammatory response syndrome (FIRS), early-onset neonatal sepsis (EONS)) in perinatal care / neonatology is steadily rising in Germany. The hands of the staff and visitors are the most important transmission vehicle of pathogens. Hence hand hygiene is one of the most important measures for the prevention of hospital infections. The different measures of hand hygiene serve to protect against the spread of contamination of the skin with obligate or potentially pathogenic pathogens. Since the use of antibiotics is generally only possible to a limited extent (especially in pregnant women and neonates in perinatal care centers) the primary prophylactic measures are of great importance.

While the importance of hand disinfection in the staff has been undisputed, there is no data on the rate of hand disinfection for visitors of perinatal care centers. Visitor at these stations are common non-compliant persons (especially children!). On the other hand, pregnant women and young mothers and newborn babies are "exposed" to a large number of visitors compared to other stations.

The investigators examine whether special measures (such as voice prompts) have a positive effect on the rate of performed hand disinfections or consecutively on the infection rate.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 7 years
* informed consent
* Member of target group: Visitor or staff

Exclusion Criteria:

* Insufficient language skills

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Total consumption of disinfectants per visitor | 9 months
  Total consumption of disinfectants per visitor (electronically counted)

SECONDARY OUTCOMES:
Prevalence of highly positive Impact tests (swab tests) | 9 months
  Prevalence of highly positive Impact tests (swab tests)
Total consumption of disinfectants (only children) per visitor | 9 months
  Total consumption of disinfectants (only children) per visitor
Infection rate of typical maternal, fetal and newborn infections | 9 months
  Infection rate of typical maternal, fetal and newborn infections

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Clinic/Perinatal Treatment Center, university hospital, Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Birnbach DJ, Nevo I, Barnes S, Fitzpatrick M, Rosen LF, Everett-Thomas R, Sanko JS, Arheart KL. Do hospital visitors wash their hands? Assessing the use of alcohol-based hand sanitizer in a hospital lobby. Am J Infect Control. 2012 May;40(4):340-3. doi: 10.1016/j.ajic.2011.05.006. Epub 2011 Aug 23. PMID 21864941
- [Background] Tromp M, Huis A, de Guchteneire I, van der Meer J, van Achterberg T, Hulscher M, Bleeker-Rovers C. The short-term and long-term effectiveness of a multidisciplinary hand hygiene improvement program. Am J Infect Control. 2012 Oct;40(8):732-6. doi: 10.1016/j.ajic.2011.09.009. Epub 2012 Jan 30. PMID 22285710
- [Background] Swoboda SM, Earsing K, Strauss K, Lane S, Lipsett PA. Isolation status and voice prompts improve hand hygiene. Am J Infect Control. 2007 Sep;35(7):470-6. doi: 10.1016/j.ajic.2006.09.009. PMID 17765560
- [Background] Huis A, van Achterberg T, de Bruin M, Grol R, Schoonhoven L, Hulscher M. A systematic review of hand hygiene improvement strategies: a behavioural approach. Implement Sci. 2012 Sep 14;7:92. doi: 10.1186/1748-5908-7-92. PMID 22978722